CLINICAL TRIAL: NCT01954381
Title: Impact of Adalimumab Therapy on Brachial Endothelial Function and Large Artery Stiffness in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-002883-26; 2011-15 (Other: AP HM)
Record Dates: First submitted 2011-10-13; First posted 2013-10-01 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2014-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Ultrasonography, Doppler; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Other)
  Interventions: Device: transthoracic echocardiographic; Device: Doppler ultrasound.; Biological: blood samples
- patient (Experimental)
  Interventions: Device: transthoracic echocardiographic; Device: Doppler ultrasound.; Biological: blood samples

INTERVENTIONS:
Device: transthoracic echocardiographic
Device: Doppler ultrasound.
Biological: blood samples

SUMMARY:
Rheumatoid arthritis (RA) is one of the most common inflammatory diseases in the general population and many cardiovascular diseases (valvular, myocardial, pericardial, coronary disease, stroke, heart failure etc.) have already been described in this disease. Large epidemiological studies have also demonstrated a higher degree of severity of atherosclerotic vascular disease in RA patients, to such a degree that several authors have highlighted the fact that, in the final analysis, the prognosis of RA is rather determined by the severity of atherosclerotic lesions.

By reducing RA-related systemic inflammation, it can therefore be hypothesized that 24 weeks of anti-TNF therapy would improve arterial endothelial function and large artery stiffness.

The proposed study will assess the effects of adalimumab therapy on these parameters. A group of 26 RA patients will be recruited from a rheumatologists association of the French PACA region (CONCERTO association). This study will be non invasive and will comprise:

* in vivo study of endothelial function by measuring the post-ischaemic dilatation by 2D ultrasound;
* study of large artery stiffness by pulse wave velocity determined by aplannation tonometry;
* study of central pulse pressure;
* evaluation of atherosclerosis-related parameters such as intima-media thickness.

The results obtained should provide a better understanding of the mechanisms involved in RA-related vascular disease and the effects of anti-TNF therapy.

In view of the high prevalence of RA, this study could potentially interest the medical community as a whole and could be largely diffused.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 years
* Patients with RA according to ACR 1987 criteria
* Indication for adalimumab therapy, according to guidelines:
* moderately to severely active RA, when the response to disease-modifying anti-rheumatic drugs, including methotrexate, is inadequate,and,severe, active and active RA in adults not previously treated with methotrexate.

Exclusion Criteria:

* Minors, pregnant women, not adequate contraception if female with childbearing potential, majors under guardianship, residents of social welfare or health care establishments, patients presenting an emergency situation, patients not covered by French social security, subjects deprived of their freedom and patients refusing to participate in the clinical research.
* Absence of informed consent
* Patients who have previously received anti-TNF therapy
* Renal failure
* History of demyelinising disease
* Any unstable medical condition
* Patients with recurrent serious infections
* History of cardiovascular or cerebrovascular disease
* History of cancer
* Patients not having TB prophylaxis as per guidelines for latent TB, or patients non-treated active tuberculosis
* Contraindication to adalimumab therapy:

  * Hypersensitivity to adalimumab or one of the excipients.
  * Active tuberculosis or other severe infections such as sepsis and opportunistic infections
  * Moderate to severe heart failure .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-10; Primary Completion 2014-10 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
evaluate the effects of 24 weeks of anti-TNF (adalimumab) therapy on | 3 YEARS
  - aortic stiffness by measuring carotid-femoral pulse wave velocity (CF-PWV)
evaluate the effects of 24 weeks of anti-TNF (adalimumab) therapy on | 3 YEARS
  - central pulse pressure (aortic)
evaluate the effects of 24 weeks of anti-TNF (adalimumab) therapy on | 3 YEARS
  - endothelial function by studying hyperaemia-induced vasodilation (FMD), reflecting the quality of endothelium-dependent vasorelaxation

SECONDARY OUTCOMES:
evaluate the resting blood pressure | 3 YEARS
evaluate the systolic pressure index | 3 YEARS
evaluate the structure of the carotid wall | 3 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique hôpitaux de Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France